CLINICAL TRIAL: NCT03390504
Title: A Phase 3 Study of Erdafitinib Compared With Vinflunine or Docetaxel or Pembrolizumab in Subjects With Advanced Urothelial Cancer and Selected FGFR Gene Aberrations
Brief Title: A Study of Erdafitinib Compared With Vinflunine or Docetaxel or Pembrolizumab in Participants With Advanced Urothelial Cancer and Selected Fibroblast Growth Factor Receptor (FGFR) Gene Aberrations
Acronym: THOR
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108401; 42756493BLC3001 (Other: Janssen Research & Development, LLC); 2017-002932-18 (EudraCT Number); 2023-510296-56-00 (Registry Identifier: EUCT number)
Expanded Access: NCT03825484 (Approved for marketing)
Record Dates: First submitted 2017-12-20; First posted 2018-01-04 (Actual); Results first posted 2025-05-14 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Urothelial Cancer
MeSH Terms: interventions — erdafitinib; vinflunine; Docetaxel; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (4):
- Cohort 1 (Arm 1A): Erdafitinib (Experimental): Participants will be screened based on Fibroblast Growth Factor Receptor Inhibitor Clinical Trial Assay (FGFRi CTA) to determine molecular eligibility and participants who meet molecular eligibility criteria will be eligible for full study screening. Participants enrolled in the study (treated with prior anti-programmed cell death protein PD-[L] 1 agent) will swallow erdafitinib tablets orally at a starting dose of 8 milligram (mg), once daily for 21 days in a 21-day cycle until disease progression, intolerable toxicity, withdrawal of consent or decision by the investigator to discontinue treatment. Dose adjustment are based on phosphate level and observed toxicity (adverse events [AEs]). Participants who enter in Long-term extension (LTE) phase will continue to receive the erdafitinib tablet as per investigator's decision.
  Interventions: Drug: Erdafitinib; Device: Fibroblast Growth Factor Receptor inhibitor Clinical Trial Assay (FGFRi CTA)
- Cohort 1 (Arm 1B): Vinflunine or Docetaxel (Experimental): Participants will be screened based on FGFRi CTA to determine molecular eligibility and participants who meet molecular eligibility criteria will be eligible for full study screening. Participants enrolled in the study (treated with prior anti-PD-[L] 1 agent) will receive vinflunine 320 milligram per meter square (mg/m^2) as a 20-minute intravenous infusion once every 3 weeks or docetaxel 75 mg/m^2 as a 1 hour intravenous infusion every 3 weeks. Treatment with either agent (choice of investigator) will be administered until disease progression, intolerable toxicity, withdrawal of consent or decision by the investigator to discontinue treatment. Dose adjustments are based on observed toxicities. Participants who enter in LTE phase will continue to receive Vinflunine or Docetaxel until the participant can commercially receive chemotherapy within the local healthcare system.
  Interventions: Drug: Vinflunine; Drug: Docetaxel; Device: Fibroblast Growth Factor Receptor inhibitor Clinical Trial Assay (FGFRi CTA)
- Cohort 2 (Arm 2A): Erdafitinib (Experimental): Participants will be screened based on FGFRi CTA to determine molecular eligibility and participants who meet molecular eligibility criteria will be eligible for full study screening. Participants enrolled in the study (no prior treatment with anti-PD-[L] 1 agent) will swallow erdafitinib tablets orally at a starting dose of 8 mg, once daily for 21 days in a 21-day cycle until disease progression, intolerable toxicity, withdrawal of consent or decision by the investigator to discontinue treatment. Dose adjustments are based on phosphate level and observed toxicity (AEs). Participants who enter in LTE phase will continue to receive the erdafitinib tablet as per investigator's decision.
  Interventions: Drug: Erdafitinib; Device: Fibroblast Growth Factor Receptor inhibitor Clinical Trial Assay (FGFRi CTA)
- Cohort 2 (Arm 2B): Pembrolizumab (Experimental): Participants will be screened based on FGFRi CTA to determine molecular eligibility and participants who meet molecular eligibility criteria will be eligible for full study screening. Participants enrolled in the study (no prior treatment with anti-PD-[L] 1 agent) will receive pembrolizumab 200 mg as a 30-minute intravenous infusion once every 3 weeks, until disease progression, intolerable toxicity, withdrawal of consent or decision by the investigator to discontinue treatment. Dose adjustments are based on observed toxicities. Participants who enter in LTE phase will continue to receive the pembrolizumab until 2 years after the first dose of pembrolizumab (at start of study) or until the participant can commercially receive pembrolizumab within the local healthcare system, whichever comes first.
  Interventions: Drug: Pembrolizumab; Device: Fibroblast Growth Factor Receptor inhibitor Clinical Trial Assay (FGFRi CTA)

INTERVENTIONS:
Drug: Erdafitinib — Participants will swallow erdafitinib tablets orally at a starting dose of 8 mg.
  Other Names: JNJ-42756493
  Arms: Cohort 1 (Arm 1A): Erdafitinib; Cohort 2 (Arm 2A): Erdafitinib
Drug: Vinflunine — Participants will receive vinflunine 320 mg/m^2 as a 20-minute intravenous infusion.
  Arms: Cohort 1 (Arm 1B): Vinflunine or Docetaxel
Drug: Docetaxel — Participants will receive docetaxel 75 mg/m^2 as a 1 hour intravenous infusion.
  Arms: Cohort 1 (Arm 1B): Vinflunine or Docetaxel
Drug: Pembrolizumab — Participants will receive pembrolizumab 200 mg as a 30-minute intravenous infusion.
  Arms: Cohort 2 (Arm 2B): Pembrolizumab
Device: Fibroblast Growth Factor Receptor inhibitor Clinical Trial Assay (FGFRi CTA) — FGFRi CTA will be used to determine molecular eligibility.

SUMMARY:
The purpose of this study is to evaluate efficacy of erdafitinib versus chemotherapy or pembrolizumab in participants with advanced urothelial cancer harboring selected fibroblast growth factor receptor (FGFR) aberrations who have progressed after 1 or 2 prior treatments, at least 1 of which includes an anti-programmed death ligand 1(PD-[L]1) agent (cohort 1) or 1 prior treatment not containing an anti-PD-(L) 1 agent (cohort 2).

DETAILED DESCRIPTION:
A study of erdafitinib versus standard of care, consisting of chemotherapy (docetaxel or vinflunine) or anti-PD-(L) 1 agent pembrolizumab, in participants with advanced urothelial cancer and selected FGFR aberrations who have progressed on or after 1 or 2 prior treatments, at least 1 of which includes an anti-PD-(L) 1 agent (cohort 1) or 1 prior treatment not containing an anti-PD-(L) 1 agent (cohort 2). It will consist of screening, treatment phase (from randomization until disease progression, intolerable toxicity, withdrawal of consent or decision by investigator to discontinue treatment, post-treatment follow-up (from end-of-treatment to participants death, withdraws consent, lost to follow-up study completion for the respective cohort, whichever comes first). The study will have long term extension (LTE) period after clinical cutoff date is achieved for final analysis of each cohort and participants eligible in the opinion of the investigator, will continue to benefit from the study intervention. Efficacy, pharmacokinetics, biomarkers, patient reported outcomes, medical resource utilization and safety will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Histologic demonstration of transitional cell carcinoma of the urothelium. Minor components ( less than [<] 50 percent [%] overall) of variant histology such as glandular or squamous differentiation, or evolution to more aggressive phenotypes such as sarcomatoid or micropapillary change are acceptable
* Metastatic or surgically unresectable urothelial cancer
* Documented progression of disease, defined as any progression that requires a change in treatment, prior to randomization
* Cohort 1: Prior treatment with an anti-PD-(L) 1 agent as monotherapy or as combination therapy; no more than 2 prior lines of systemic treatment. Cohort 2: No prior treatment with an anti-PD-(L) 1 agent; only 1 line of prior systemic treatment. Subjects who received neoadjuvant or adjuvant chemotherapy and showed disease progression within 12 months of the last dose are considered to have received systemic therapy in the metastatic setting.
* A woman of childbearing potential who is sexually active must have a negative pregnancy test (beta human chorionic gonadotropin [beta hCG]) at Screening (urine or serum)
* Participants must meet appropriate molecular eligibility criteria
* Eastern Cooperative Oncology Group (ECOG) performance status Grade 0, 1, or 2
* Adequate bone marrow, liver, and renal function

Exclusion Criteria:

* Treatment with any other investigational agent or participation in another clinical study with therapeutic intent within 30 days prior to randomization
* Active malignancies (that is, requiring treatment change in the last 24 months). The only allowed exceptions are: urothelial cancer, skin cancer treated within the last 24 months that is considered completely cured, localized prostate cancer with a gleason score of 6 (treated within the last 24 months or untreated and under surveillance) and localized prostate cancer with a gleason score of 3+4 that has been treated more than 6 months prior to full study screening and considered to have a very low risk of recurrence.
* Symptomatic central nervous system metastases
* Received prior fibroblast growth factor receptor (FGFR) inhibitor treatment
* Known allergies, hypersensitivity, or intolerance to erdafitinib or its excipients
* Current central serous retinopathy (CSR) or retinal pigment epithelial detachment of any grade.
* History of uncontrolled cardiovascular disease
* Impaired wound healing capacity defined as skin/decubitus ulcers, chronic leg ulcers, known gastric ulcers, or unhealed incisions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 629 (Actual)
Dates: Start 2018-03-23 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2026-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (345):
- United States (26):
  - Alaska Urological Institute dba Alaska Clinical Research Center, Anchorage, Alaska
  - University of Calif Davis Medical Center, Sacramento, California
  - St. Helena Hospital - Martin-O'Neil Cancer Center, St. Helena, California
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - University of Miami Sylvester Cancer Center, Miami, Florida
  - Mid Florida Hematology Oncology, Orange, Florida
  - Piedmont Cancer Institute, Atlanta, Georgia
  - Rush University, Chicago, Illinois
  - Edward Hines Jr V A Hospital, Hines, Illinois
  - Norton Cancer Institute, Louisville, Kentucky
  - Maryland Oncology Hematology, PA, Lanham, Maryland
  - University of Michigan Health System, Ann Arbor, Michigan
  - VA Sierra Nevada Health Care System, Reno, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Weill Cornell Medical College, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Levine Cancer Institute, Carolinas HealthCare System, Charlotte, North Carolina
  - W G Bill Hefner VA Medical Center, Salisbury, North Carolina
  - Oncology Hematology Care, Cincinnati, Ohio
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas
  - Texas Oncology-Memorial City, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Texas Oncology Tyler, Tyler, Texas
  - INOVA Dwiight &Martha Schar Cancer Institute, Fairfax, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - VA Puget Sound Healthcare System, Seattle, Washington
- Argentina (8):
  - Sociedade Beneficente de Senhoras Hospital Sirio Libanes, Buenos Aires
  - Centro Oncológico Korben, Buenos Aires
  - CEMIC Saavedra, Buenos Aires
  - Cemaic Centro Privado de Especialidades Medicas Ambulatorias e Investigacion Clinica, Córdoba
  - Centro Urologico Profesor Bengio, Córdoba
  - Hospital Privado de Comunidad, Mar del Plata
  - Centro de Investigacion Pergamino SA, Pergamino
  - Clínica Viedma, Viedma
- Australia (6):
  - Chris O'Brien Lifehouse, Camperdown
  - Peninsula & South Eastern Haematology and Oncology Group, Frankston
  - St George Hospital, Kogarah
  - Peter MacCallum Cancer Centre, Melbourne
  - Frankston Hospital, Melbourne
  - Fiona Stanley Hospital, Murdoch
- Austria (5):
  - LKH-Univ. Klinikum Graz, Graz
  - Ordensklinikum Linz GmbH Elisabethinen, Linz
  - LKH - Universitätsklinikum der PMU Salzburg, Salzburg
  - Krankenhaus der Barmherzigen Brüder, Vienna
  - Medical University Vienna MUV, Vienna
- Belgium (9):
  - OLV Ziekenhuis Aalst, Aalst
  - ZNA Middelheim, Antwerp
  - Cliniques Universitaires Saint Luc, Brussels
  - Clinique Notre Dame de Grâce, Charleroi
  - AZ Maria Middelares, Ghent
  - UZ Gent, Ghent
  - CHC MontLegia, Liège
  - Sint-Augustinus AZ, Wilrijk
  - CHU UCL Namur - Site Godinne, Yvoir
- Brazil (22):
  - Fundacao Pio XII, Barretos
  - Universidade Federal De Minas Gerais - Hospital das Clínicas, Belo Horizonte
  - Nucleo de Ensino e Pesquisa do Instituto Mario Penna, Belo Horizonte
  - Instituto de Oncologia do Parana, Curitiba
  - Liga Paranaense de Combate ao Cancer, Curitiba
  - Associacao de Combate ao Cancer em Goias - Hospital de Cancer Araujo Jorge, Goiânia
  - Clínica de Neoplasias Litoral Ltda., Itajaí
  - Fundacao Doutor Amaral Carvalho, Jaú
  - Liga Norte Riograndense Contra O Cancer, Natal
  - Hospital das Clinicas de Porto Alegre, Porto Alegre
  - Hospital Nossa Senhora da Conceicao S A, Porto Alegre
  - Ministerio da Saude Instituto Nacional do Cancer, Rio de Janeiro
  - Oncoclinicas Rio de Janeiro S A, Rio de Janeiro
  - Hospital Sao Rafael, Salvador
  - CEPHO Centro de Estudos e Pesquisa de Hematologia e Oncologia, Santo André
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto Hospital de Base, São José do Rio Preto
  - Sociedade Beneficente de Senhoras Hospital Sirio Libanes, São Paulo
  - Fundacao Antonio Prudente A C Camargo Cancer Center, São Paulo
  - Instituto Brasileiro de Controle do Cancer - Sao Camilo Oncologia, São Paulo
  - Instituto D Or de Pesquisa e Ensino IDOR, São Paulo
  - Sociedade Beneficente Israelita Brasileira Hospital Albert Einstein, São Paulo
  - Instituto de Oncologia de Sorocaba Onco Clinicas Especializadas, Sorocaba
- Bulgaria (5):
  - UMHAT 'Dr. Georgi Stranski', EAD, Pleven
  - Complex Oncology Center - Plovdiv EOOD, Plovdiv
  - Multiprofile Hospital for Active Treatment 'Tokuda Hospital Sofia', Sofia
  - UMHAT Sofia Med, Sofia
  - Multiprofile Hospital for Active Treatment 'Sveta Marina' EAD, Varna
- Canada (6):
  - BC Cancer Agency - Southern Interior, Kelowna, British Columbia
  - Vancouver Cancer Centre, Vancouver, British Columbia
  - Cancercare Manitoba, Winnipeg, Manitoba
  - Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario
  - Princess Margaret Hospital- UHN, Toronto, Ontario
  - Saskatchewan Cancer Agency (SCA) - Allan Blair Cancer Centre, Regina, Saskatchewan
- China (24):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing
  - Peking University First Hospital, Beijing
  - Beijing Friendship Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - Beijing Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - The First Bethune Hospital of Jilin University, Changchun
  - Sichuan Provincial Peoples Hospital, Chengdu
  - Sichuan University Huaxi Hospital, Chengdu
  - Chongqing University Cancer Hospital, Chongqing
  - Sun Yat Sen University Cancer Center, Guangzhou
  - Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou
  - Guangzhou First Municipal People's Hospital, Guangzhou
  - Zhejiang Provincial People's Hospital, Hangzhou
  - Sir Run Run Shaw Hospital Zhejiang University School of Medicine, Hangzhou
  - The First Affliated Hospital Of Nanchang University, Nanchang
  - Nanjing Drum Tower Hospital, Nanjing
  - Jiangsu Cancer Hospital, Nanjing
  - Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - Huadong Hospital Affiliated to Fudan University, Shanghai
  - Shengjing Hospital Of China Medical University, Shenyang
  - Shenzhen university General Hospital, Shenzhen
  - First Affiliated Hospital Of Wenzhou Medical College, Wenzhou
  - The First Affiliated Hospital of Xian Jiaotong University, Xi'an
- France (24):
  - Institut de Cancerologie de l Ouest ICO, Angers
  - Hopital Jean Minjoz, Besançon
  - Institut Bergonie, Bordeaux
  - CHRU Brest - Hopital Morvan, Brest
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Georges-François Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Hôpital Privé Le Bois, Lille
  - Groupe Hospitalier Bretagne Sud, Lorient
  - Hopital de la Timone, Marseille
  - Institut Regional du Cancer de Montpellier Val d'Aurelle, Montpellier
  - Centre Antoine Lacassagne, Nice
  - Institut de Cancérologie du Gard, Nîmes
  - Hopital Europeen Georges-Pompidou, Paris
  - Hospital Saint-Louis, Paris
  - Hospices Civils de Lyon HCL, Pierre-Bénite
  - CHU De Poitiers, Poitiers
  - Centre Eugene Marquis, Rennes
  - Centre de radiothérapie et d'Oncologie médicale de l'Essonne, Ris-Orangis
  - Institut de Cancérologie de Loire, Saint-Priest-en-Jarez
  - Hôpitaux Universitaires de Strasbourg - Hôpital de Hautepierre, Strasbourg
  - Institut Claudius Regaud, Toulouse
  - Centre Les Dentellieres, Valenciennes
  - Institut Gustave Roussy, Villejuif
- Germany (19):
  - Vivantes Klinikum Am Urban, Berlin
  - Stadtisches Klinikum Braunschweig gGmbH-Klinik fur Urologie und Uroonkologie, Braunschweig
  - Universitatsklinikum Carl Gustav Carcus Dresden, Dresden
  - Universitaetsklinikum Duesseldorf, Düsseldorf
  - Friedrich-Alexander Universitaet Urologische Universitaetskl, Erlangen
  - Universitatsklinikum Frankfurt, Frankfurt
  - Universitatsklinikum Freiburg, Freiburg im Breisgau
  - Universitatsmedizin Gottingen, Göttingen
  - Universitätsmedizin Greifswald, Greifswald
  - Asklepios Klinik Altona, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitatsklinikum Schleswig Holstein Campus Lubeck, Lübeck
  - Medizinische Fakultät Mannheim der Universität Heidelberg, Mannheim
  - Universitaetsklinikum Muenster, Münster
  - Studienpraxis Urologie Drs. Feyerabend, Nürtingen
  - Caritas-Krankenhaus St. Josef, Regensburg
  - Universitaetsmedizin Rostock, Rostock
  - MVZ-Onkologie Velbert GbR, Velbert
  - Kliniken Nordoberpfalz AG/Klinikum Weiden, Weiden
- Greece (9):
  - University of Athens Medical School - Regional General Hospi, Athens
  - Errikos Dunant Hospital Center, Athens
  - Athens Medical Center, Athens
  - Metropolitan General A E, Athens
  - University Hospital Of Larissa, Larissa
  - University General Hospital of Rio Patras, Pátrai
  - Interbalkan European Medical Center, Thessaloniki
  - Euromedica General Clinic, Thessaloniki
  - Papageorgiou General Hospital Of Thessaloniki, Thessaloniki
- Hungary (5):
  - Semmelweis Egyetem, Budapest
  - Országos Onkológiai Intézet, Urogenitális Tumorok és Klinikai Farmakológiai Osztály, Budapest
  - Budapesti Uzsoki Utcai Korhaz, Budapest
  - Szabolcs-Szatmar-Bereg Megyei Korhazak es Egyetemi Oktatokorhaz, Nyíregyháza
  - Pecsi Tudomanyegyetem Klinikai Kozpont, Pécs
- Israel (7):
  - Rambam Health Care Campus, Haifa
  - Hadassah Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Beilinson Hospital, Petach Tikvah
  - Sourasky Medical Center, Tel Aviv
  - The Chaim Sheba Medical Center, Tel Litwinsky
  - Assaf Harofeh Medical Center, Tzrifin
- Italy (27):
  - Azienda Ospedaliera Nazionale SS. Antonio e Biagio e Cesare Arrigo Alessandria, Alessandria
  - Ospedale S. Donato - Asl 8 Arezzo, Arezzo
  - CRO IRCCS Istituto Nazionale Tumori, Aviano
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia Presidio Spedali Civili, Brescia
  - Istituti Ospitalieri di Cremona, AO di Cremona, Cremona
  - Oncologia Medica, Florence
  - SPDC Villa Scassi, Genova
  - UOC Oncologia Ospedale Provinciale di Macerata, Macerata
  - IRST Meldola Forli, Meldola
  - IRCCS Ospedale San Raffaele, Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - European Institute of Oncology, Milan
  - AOU Policlinico di Modena, Modena
  - IRCCS-Fondazione Pascale, Napoli
  - Ospedale Maggiore della Carita, Novara
  - Aou San Luigi Gonzaga, Orbassano
  - Istituto Oncologico Veneto Iov Irccs Padova, Padua
  - AOU di Parma, Parma
  - IRCCS Policlinico San Matteo, Pavia
  - Ist. Clinici Scientifici Maugeri - Unità Operativa di Oncolo, Pavia
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Usl 7 Siena - Ospedale Alta Valdelsa ASL TOSCANA SUD-EST, Poggibonsi (SI)
  - Fondazione Policlinico Universitario A Gemelli IRCCS, Roma
  - Azienda Ospedaliera Universitaria Senese Policlinico Santa Maria alle Scotte, Siena
  - Oncologia Medica-Città Della Salute E Della Scienza Di Torino, Torino
  - Azienda Ospedaliero - Universitaria Ospedali Riuniti, Torrette Di Ancona
- Japan (23):
  - Chiba Cancer Center, Chiba
  - Hirosaki University Hospital, Hirosaki
  - National Cancer Center Hospital East, Kashiwa
  - Kagawa University Hospital, Kita Gun
  - Kobe City Medical Center General Hospital, Kobe
  - Dokkyo Medical University Saitama Medical Center, Koshigaya
  - Aso Co.,Ltd Iizuka Hospital, Matsuyama
  - University of Miyazaki Hospital, Miyazaki
  - Nagano Municipal Hospital, Nagano
  - Aichi Cancer Center Hospital, Nagoya
  - Osaka International Cancer Institute, Osaka
  - Osaka City University Hospital, Osaka
  - Kindai University Hospital, Ōsaka-sayama
  - Gunma Prefectural Cancer Center, Ōta-ku
  - Kitasato University Hospital, Sagamihara
  - Toho University Sakura Medical Center, Sakura
  - National Hospital Organization Hokkaido Cancer Center, Sapporo
  - Tokyo Women's Medical University Hospital, Shinjuku-ku
  - Toranomon Hospital, Tokyo
  - The Cancer Institute Hospital of JFCR, Tokyo
  - University of Tsukuba Hospital, Tsukuba
  - Yamaguchi University Hospital, Ube
  - Yokohama City University Medical Center, Yokohama
- Mexico (3):
  - Medicos Especialistas en Cancer, S.C., Aguascalientes
  - Centro Estatal de Cancerología de Chihuahua, Chihuahua City
  - Oncologia Integral Satelite, Naucalpan
- Netherlands (3):
  - Antoni van Leeuwenhoek, Amsterdam
  - St. Antonius Ziekenhuis Nieuwegein, Nieuwegein
  - Haga ziekenhuis, The Hague
- Poland (4):
  - Centrum Onkologii im Prof F Lukaszczyka w Bydgoszczy, Bydgoszcz
  - Centralny Szpital Kliniczny MSWiA w Warszawie, Warsaw
  - Narodowy Instytut Onkologii im Marii Sklodowskiej Curie Panstwowy Instytut Badawczy, Warsaw
  - Uniwersytecki Szpital Kliniczny we Wroclawiu, Wroclaw
- Portugal (5):
  - Champalimaud Foundation Champalimaud Centre, Lisbon
  - Hospital Lusíadas, Lisbon
  - H. Santa Maria - Centro Hospitalar de Lisboa Norte, Lisbon
  - Uls Sao Jose - Hosp. Sto Antonio Dos Capuchos, Lisbon
  - Instituto Portugues de Oncologia, Porto
- Russia (28):
  - Altai Regional Oncology Dispensary, Barnaul
  - Chelyabinsk Regional Clinical Center Of Oncology And Nuclear Medicine, Chelyabinsk
  - Irkutsk Regional Oncology Dispensary, Irkutsk
  - Ivanovo Regional Oncology Dispensary, Ivanovo
  - Kostroma regional oncology dispensary, Kostroma
  - Leningrad Regional Oncology Dispensary, Kuzmolovsky
  - City Clinical Hospital n.a. D.D.Pletnev, Moscow
  - FSBSI 'N. N. Blokhin Russian Cancer Research Center', Moscow
  - Russian Scientific Center of Roentgenoradiology, Moscow
  - I.M. Sechenov First Moscow State Medical University, Moscow
  - Hertzen Oncology Research Institute, Moscow
  - City Clinical Hospital #1, Nal'chik
  - Privolzhsky District Medical Center under the Federal Medico-Biological Agency, Nizhny Novgorod
  - Clinical Oncology Dispensary, Omsk
  - GBUZ of Stavropol region Pyatigorsk Oncological Dispensary, Pyatigorsk
  - LLC 'Strategic Medical Systems', Saint Petersburg
  - Clinical hopital n/a Petra velikogo, Saint Petersburg
  - Private Medical Institution Euromedservice, Saint Petersburg
  - Pavlov First Saint Petersburg State Medical University, Saint Petersburg
  - Russian Scientific Center of Radiology and Surgical Technologies, Saint Petersburg
  - Saint-Petersburg Clinical Scientific And Practical Center For Special Types Of Medical Care, Saint Petersburg
  - FGBOU Vo Mordovian National Research State University N. A. N.P. Ogareva, Saransk
  - Saratov State Medical University, Saratov
  - LLC Uromed, Smolensk
  - GBUZ Oncology Centre #2 of Healthcare Department of Krasno, Sochi
  - Multifunctional clinical medical center 'Medical city', Tyumen
  - Bashkiria State Medical University, Ufa
  - Vologda Regional Oncological Dispensary, Vologda
- South Korea (12):
  - Pusan National University Hospital, Busan
  - Chungnam National University Hospital, Daejeon
  - National Cancer Center, Goyang-si
  - Chonnam National University Hospital, Gwangju
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - Yonsei University Wonju Severance Christian Hospital, Wŏnju
- Spain (20):
  - Hosp. Univ. Infanta Cristina, Badajoz
  - Institut Català D'Oncologia-Hospital Universitari Germans Trias I Pujol, Badalona
  - Hosp Clinic de Barcelona, Barcelona
  - Hosp. de La Santa Creu I Sant Pau, Barcelona
  - Hosp. San Pedro de Alcantara, Cáceres
  - Hosp Reina Sofia, Córdoba
  - Hosp. Univ. Virgen de Las Nieves, Granada
  - Complejo Hospitalario de Jaen, Jaén
  - Hosp. Univ. Insular de Gran Canaria, Las Palmas de Gran Canaria
  - Hosp. Univ. Lucus Augusti, Lugo
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Univ. La Paz, Madrid
  - Hosp. Univ. Pta. de Hierro Majadahonda, Majadahonda
  - ALTHAIA, Xarxa Assistencial Universitària de Manresa, Manresa
  - Hosp. de Navarra, Pamplona
  - Hosp. Virgen Macarena, Seville
  - Hosp. Virgen Del Rocio, Seville
  - Hosp. Gral. Univ. Valencia, Valencia
  - Hosp. Univ. I Politecni La Fe, Valencia
  - Hosp. Univ. Miguel Servet, Zaragoza
- Taiwan (11):
  - Kaohsiung Medical University Chung Ho Memorial Hospital, Kaohsiung City
  - Chang Gung Medical Foundation, Niao-Sung Hsiang
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Chi Mei Medical Center Yong Kang, Tainan
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center, Taipei
  - Chang-Gung Memorial Hospital, LinKou Branch, Taoyuan District
- Turkey (Türkiye) (12):
  - Baskent University Adana Practice and Research Center Kisla Health Campus, Adana
  - Hacettepe University Medical Faculty, Ankara
  - Bezmialem University Medical Faculty, Istanbul
  - Istanbul University Cerrahpasa Medical Faculty, Istanbul
  - Bakirkoy Training and Research Hospital, Istanbul
  - Medipol Mega University Hospital, Istanbul
  - T C Saglik Bakanlıgi Goztepe Prof Dr Suleyman Yalcın Sehir Hastanesi, Istanbul
  - Pendik Training and Research Hospital, Istanbul
  - Ege University, Izmir
  - Dokuz Eylul Universitesi Tip Fakultesi, Izmir
  - Kocaeli University Medical Faculty, Kocaeli
  - Inonu Universitesi Turgut Ozal Tip Merkezi, Ic Hastaliklari, Malatya
- Ukraine (13):
  - Municipal Institution 'Clinical Oncology Dispensary' Under Dnipropetrovsk Regional Council, Dnipro
  - Dnipropetrovsk State Medical Academy, Dnipropetrovsk City Multifield Clinical Hospital # 4, Dnipro
  - MI Dnipropetrovsk Region Clinical Hospital n a I.I.Mechnikov, Dnipropetrovsk
  - Ivano-Frankivsk Regional Clinical Hospital, Ivano-Frankivsk
  - Regional Medical Clinical Center for Urology and Nephrology named after V.I. Shapoval, Kharkiv
  - Municipal non-profit enterprise 'Regional Center of Oncology', Kharkiv
  - National Cancer Institute, Kyiv
  - State Institution Institute of Urology NAMS of Ukraine based on Kyiv City Clinical Oncology Center, Kyiv
  - Communal Noncommercial Enterprise of Lviv Regional Council 'Lviv Regional Clinical Hospital', Lviv
  - Transkarpathian Regional University Oncology Clinic, Uzhhorod
  - Podilskiy Regional Center of Oncology, Vinnitsa
  - Zaokod, Zaporizhzhia
  - Zaporizhzhia medical Academy of postgraduate education, Zaporizhzhia Regoinal Clinical Hospital, Zaporizhzhia
- United Kingdom (9):
  - University Hospitals Bristol - Bristol Haematology & Oncolog, Bristol
  - St Bartholomew's Hospital, London
  - Sarah Cannon Research Institute, London
  - Charing Cross Hospital, London
  - The Christie NHS Foundation Trust Christie Hospital, Manchester
  - Derriford Hospital-Department of Medical Oncology, Plymouth
  - University of Sheffield, Sheffield
  - Southampton General Hospital, Southampton
  - Royal Marsden Hospital, Sutton

REFERENCES:
- [Derived] Loriot Y, Matsubara N, Park SH, Huddart RA, Burgess EF, Houede N, Banek S, Guadalupi V, Ku JH, Valderrama BP, Tran B, Triantos S, Kean Y, Akapame S, Deprince K, Mukhopadhyay S, Stone NL, Siefker-Radtke AO; THOR Cohort 1 Investigators. Erdafitinib or Chemotherapy in Advanced or Metastatic Urothelial Carcinoma. N Engl J Med. 2023 Nov 23;389(21):1961-1971. doi: 10.1056/NEJMoa2308849. Epub 2023 Oct 21. PMID 37870920

RESULTS

PARTICIPANT FLOW:
Recruitment Details: With the implementation of Protocol Amendment 6 (20 January 2023), long term extension (LTE) phase was added in the study.
Groups:
- Cohort 1: Arm 1A: Erdafitinib 8 mg/9 mg: Participants with advanced urothelial cancer and selected fibroblast growth factor receptor (FGFR) aberrations who were previously treated with anti-programmed death-ligand 1 (PD-[L]1) agent were randomized to receive erdafitinib tablet orally once daily starting from Day 1 through Day 21 in each subsequent 21-day cycles starting from Cycle 1 until disease progression, intolerable toxicity, withdrawal of consent, decision by the investigator to discontinue treatment or end of treatment. All subjects randomized to erdafitinib received erdafitinib 8 mg once daily from Day 1 to Day 14 of Cycle 1. On Day 14 of Cycle 1, serum phosphate concentration was measured. Based on the measured serum phosphate levels the treatment could be up-titrated to erdafitinib 9 mg. With the implementation of Protocol Amendment 6 (20 January 2023), participants who benefited from the study drug as determined by investigator, continued to receive study drug in the LTE phase. The participants who did not enter LTE phase discontinued the study.
- Cohort 1: Arm 1B: Chemotherapy (Vinflunine 320 mg/m^2 or Docetaxel 75 mg/m^2): Participants with advanced urothelial cancer and selected FGFR aberrations who were previously treated with PD-(L)1 agent were randomized to receive chemotherapy (vinflunine 320 milligrams per meter square [mg/m^2] intravenous [IV] infusion or docetaxel 75 mg/m^2 IV infusion) on Day 1 of every cycle (each cycle 21 days) until disease progression, intolerable toxicity, withdrawal of consent or decision by the investigator to discontinue treatment or end of treatment. The choice of chemotherapy regimen at each site was determined by the investigator. Participants were then followed up for safety until death, withdrawal of consent, loss of follow up or end of study. With the implementation of Protocol Amendment 6 (20 January 2023), participants who benefited from the study drug as determined by investigator, continued to receive study drug in the LTE phase. The participants who did not enter LTE phase discontinued the study.
- Cohort 2: Arm 2A: Erdafitinib 8 mg/ 9 mg: Participants with advanced urothelial cancer and selected FGFR aberrations who were not previously treated with anti-PD-(L)1 agent were randomized to receive erdafitinib tablet orally once daily starting from Day 1 through Day 21 in each subsequent 21-day cycles starting from Cycle 1 until disease progression, intolerable toxicity, withdrawal of consent, decision by the investigator to discontinue treatment or end of treatment. All subjects randomized to erdafitinib received erdafitinib 8 mg once daily from Day 1 to Day 14 of Cycle 1. On Day 14 of Cycle 1, serum phosphate concentration was measured. Based on the measured serum phosphate levels the treatment could be up-titrated to erdafitinib 9 mg. With the implementation of Protocol Amendment 6 (20 January 2023), participants who benefited from the study drug as determined by investigator, continued to receive study drug in the LTE phase. The participants who did not enter LTE phase discontinued the study.
- Cohort 2: Arm 2B: Pembrolizumab 200 mg: Participants with advanced urothelial cancer and selected FGFR aberrations who were not previously treated with PD-(L)1 agent were randomized to receive pembrolizumab 200 mg IV infusion on Day 1 of every cycle (each cycle 21 days) until disease progression, intolerable toxicity, withdrawal of consent, or decision by the investigator to discontinue treatment or end of treatment. Participants were then followed up for safety until death, withdrawal of consent, loss of follow up or end of study. With the implementation of Protocol Amendment 6 (20 January 2023), participants who benefited from the study drug as determined by investigator, continued to receive study drug in the LTE phase. The participants who did not enter LTE phase discontinued the study.
Period: Overall Study
Arm/Group | Cohort 1: Arm 1A: Erdafitinib 8 mg/9 mg | Cohort 1: Arm 1B: Chemotherapy (Vinflunine 320 mg/m^2 or Docetaxel 75 mg/m^2) | Cohort 2: Arm 2A: Erdafitinib 8 mg/ 9 mg | Cohort 2: Arm 2B: Pembrolizumab 200 mg
Started | 143 | 135 | 175 | 176
Treated | 142 | 117 | 173 | 173
Completed (Participants who died were considered to have completed the study as per protocol.) | 137 | 114 | 168 | 167
Not Completed | 6 | 21 | 7 | 9
Not completed — Lost to Follow-up | 2 | 4 | 0 | 1
Not completed — Withdrawal by Subject | 3 | 15 | 5 | 2
Not completed — Other | 1 | 2 | 2 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Arm 1A: Erdafitinib 8 mg/9 mg | Cohort 1: Arm 1B: Chemotherapy (Vinflunine 320 mg/m^2 or Docetaxel 75 mg/m^2) | Cohort 2: Arm 2A: Erdafitinib 8 mg/ 9 mg | Cohort 2: Arm 2B: Pembrolizumab 200 mg | Total
Number analyzed (Participants) | 143 | 135 | 175 | 176 | 629
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 61 | 47 | 67 | 70 | 245
  >=65 years | 82 | 88 | 108 | 106 | 384
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.0 (10.23) | 67.9 (9.07) | 67.0 (8.49) | 65.9 (10.20) | 66.4 (9.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 38 | 33 | 44 | 158
  Male | 100 | 97 | 142 | 132 | 471
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 5 | 5 | 17
  Not Hispanic or Latino | 119 | 100 | 126 | 139 | 484
  Unknown or Not Reported | 21 | 31 | 44 | 32 | 128
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 39 | 42 | 37 | 36 | 154
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 4 | 0 | 5
  White | 85 | 66 | 95 | 111 | 357
  More than one race | 0 | 1 | 0 | 1 | 2
  Unknown or Not Reported | 19 | 25 | 39 | 28 | 111
Region of Enrollment [Count of Participants; unit: Participants]
  ARGENTINA | 1 | 1 | 0 | 0 | 2
  AUSTRALIA | 6 | 2 | 1 | 5 | 14
  AUSTRIA | 2 | 2 | 2 | 2 | 8
  BELGIUM | 5 | 2 | 6 | 2 | 15
  BRAZIL | 4 | 3 | 11 | 11 | 29
  CANADA | 2 | 0 | 2 | 4 | 8
  CHINA | 8 | 11 | 10 | 15 | 44
  FRANCE | 20 | 28 | 34 | 25 | 107
  GERMANY | 6 | 10 | 1 | 9 | 26
  GREECE | 4 | 4 | 6 | 5 | 19
  HUNGARY | 2 | 1 | 1 | 2 | 6
  ISRAEL | 2 | 3 | 1 | 1 | 7
  ITALY | 14 | 11 | 15 | 15 | 55
  JAPAN | 15 | 15 | 11 | 10 | 51
  NETHERLANDS | 4 | 0 | 1 | 0 | 5
  POLAND | 0 | 0 | 1 | 0 | 1
  PORTUGAL | 0 | 0 | 4 | 1 | 5
  RUSSIAN FEDERATION | 2 | 2 | 7 | 9 | 20
  SOUTH KOREA | 12 | 13 | 10 | 6 | 41
  SPAIN | 14 | 12 | 15 | 16 | 57
  TAIWAN | 4 | 2 | 6 | 4 | 16
  TURKEY | 3 | 1 | 13 | 19 | 36
  UKRAINE | 0 | 0 | 9 | 7 | 16
  UNITED KINGDOM | 6 | 7 | 2 | 6 | 21
  UNITED STATES | 6 | 5 | 6 | 2 | 19
  Bulgaria | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall survival was measured from the date of randomization to the date of the participant's death.
Time Frame: From randomization (3 days prior to Cycle 1 Day 1) until death due to any cause (maximum up to 51.7 months)
Population: Intent-to-Treat (ITT) analysis set included all randomized participants. Participants in this population were analyzed according to the treatment to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1: Arm 1A: Erdafitinib 8 mg/9 mg | Cohort 1: Arm 1B: Chemotherapy (Vinflunine 320 mg/m^2 or Docetaxel 75 mg/m^2) | Cohort 2: Arm 2A: Erdafitinib 8 mg/ 9 mg | Cohort 2: Arm 2B: Pembrolizumab 200 mg
Number analyzed (Participants) | 143 | 135 | 175 | 176
Months | 12.06 [10.25 to 16.36] | 8.74 [6.67 to 10.71] | 10.91 [9.23 to 12.58] | 11.07 [9.72 to 13.63]
Statistical Analysis 1: Comparison: Cohort 1: Arm 1A: Erdafitinib 8 mg/9 mg vs Cohort 1: Arm 1B: Chemotherapy (Vinflunine 320 mg/m^2 or Docetaxel 75 mg/m^2); Test type: Superiority; p = 0.0031, Log Rank; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.48 to 0.86]
Statistical Analysis 2: Comparison: Cohort 2: Arm 2A: Erdafitinib 8 mg/ 9 mg vs Cohort 2: Arm 2B: Pembrolizumab 200 mg; Test type: Superiority; p = 0.2121, Stratified log-rank test; Hazard Ratio (HR) = 1.16, 95% CI 2-sided [0.92 to 1.48]

2. Secondary Outcome: Progression Free Survival (PFS) as Per Response Evaluation Criteria in Solid Tumors (RECIST) Version (v) 1.1
Description: PFS was defined as the time from the date of randomization to the date of disease progression or relapse from complete response (CR) based on investigator assessment using RECIST v 1.1, or death due to any cause, whichever occurred first. As per RECIST v 1.1, CR was defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must had reduction in the short axis to less than (<) 10 millimeters (mm). Progressive disease (PD) was defined as at least 20 percent (%) increase in the sum of diameters of measured lesions taking as references the smallest sum of diameters recorded on study (including baseline) and an absolute increase of greater than or equal to (>=) 5 mm or appearance of at least 1 new lesion.
Time Frame: From randomization (3 days prior to Cycle 1 Day 1) until disease progression or relapse from CR or death (maximum up to 51.7 months)
Population: ITT analysis set included all randomized participants. Participants in this population were analyzed according to the treatment to which they were randomized. Here 'N' (overall number of participants analyzed) refers to the number of participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1: Arm 1A: Erdafitinib 8 mg/9 mg | Cohort 1: Arm 1B: Chemotherapy (Vinflunine 320 mg/m^2 or Docetaxel 75 mg/m^2) | Cohort 2: Arm 2A: Erdafitinib 8 mg/ 9 mg | Cohort 2: Arm 2B: Pembrolizumab 200 mg
Number analyzed (Participants) | 115 | 103 | 156 | 158
Months | 5.39 [4.37 to 5.62] | 2.73 [2.10 to 4.17] | 4.44 [4.07 to 5.49] | 2.69 [1.64 to 3.02]

3. Secondary Outcome: Objective Response Rate (ORR) Per RECIST Version 1.1
Description: ORR was defined as the percentage of participants who achieved CR or partial response (PR) as determined by investigator per RECIST v1.1. CR was defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must had reduction in the short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From start of the treatment (Day 1 Cycle 1) up to maximum of 51.7 months
Population: ITT analysis set included all randomized participants. Participants in this population were analyzed according to the treatment to which they were randomized.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1: Arm 1A: Erdafitinib 8 mg/9 mg | Cohort 1: Arm 1B: Chemotherapy (Vinflunine 320 mg/m^2 or Docetaxel 75 mg/m^2) | Cohort 2: Arm 2A: Erdafitinib 8 mg/ 9 mg | Cohort 2: Arm 2B: Pembrolizumab 200 mg
Number analyzed (Participants) | 143 | 135 | 175 | 176
Percentage of participants | 46.9 | 12.6 | 40.0 | 21.6

4. Secondary Outcome: Change From Baseline in Physical Functioning Scales of the Functional Assessment of Cancer Therapy - Bladder Cancer (FACT-Bl)
Description: The FACT-Bl consisted of 39 items, with 5-point Likert scales, covering 5 primary domains: physical well-being, social/family well-being, emotional well-being, functional well-being and additional concerns for participants with bladder cancer. The response options ranged from 0 to 4 where, 0='Not at all" and 4= "very much." FACT-Bl total score ranged from 0 (worst) to 156 (best). The higher the score, the better the quality of life (QOL). The baseline value was defined as the value collected at the time closest to but prior to the randomization.
Time Frame: Baseline up to Cycle 11 (each cycle was of 21 days)
Population: Analysis population set included in ITT (all randomized) participants with available data for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Cohort 1: Arm 1A: Erdafitinib 8 mg/9 mg | Cohort 1: Arm 1B: Chemotherapy (Vinflunine 320 mg/m^2 or Docetaxel 75 mg/m^2) | Cohort 2: Arm 2A: Erdafitinib 8 mg/ 9 mg | Cohort 2: Arm 2B: Pembrolizumab 200 mg
Number analyzed (Participants) | 136 | 130 | 175 | 176
Score on scale | -3.70 (2.365) | -5.28 (2.746) | -4.56 (1.946) | -0.26 (1.980)

5. Secondary Outcome: Time Until Symptom Deterioration
Description: Time until symptom deterioration was defined as the first time to increase in urinary bladder cancer symptoms score from the day of randomization beyond a meaningful change threshold compared to baseline. The urinary bladder cancer symptom score was subset of FACT-Bl which included 3 items related to urinary symptoms, 5-point Likert scale. Response options ranged from 0 to 4, 0 = Not at all, 1= A little bit, 2= Somewhat, 3=Quite a bit, 4 = Very much. A response of 0 indicated no symptoms and 4 indicated severe symptoms. Total sum scores ranged from 0 to 12, higher scores indicate relatively poor quality of life.
Time Frame: Randomization (3 days prior to Cycle 1 Day 1) up to maximum of 51.7 months
Population: Analysis population set included in ITT (all randomized) participants with available data for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1: Arm 1A: Erdafitinib 8 mg/9 mg | Cohort 1: Arm 1B: Chemotherapy (Vinflunine 320 mg/m^2 or Docetaxel 75 mg/m^2) | Cohort 2: Arm 2A: Erdafitinib 8 mg/ 9 mg | Cohort 2: Arm 2B: Pembrolizumab 200 mg
Number analyzed (Participants) | 136 | 130 | 175 | 176
Months | 1.5 [0.82 to 2.83] | 2.8 [1.51 to 5.32] | 2.1 [1.41 to 3.48] | 2.1 [1.38 to 4.17]

6. Secondary Outcome: Percentage of Participants With Shift From Baseline in Patient-Global Impression of Severity (PGIS)
Description: The PGI-S was a single item patient-reported measure assessing participants' impression of severity in bladder cancer symptoms. It uses a 4-point Likert scale as follows: symptoms are: 0-"absent (no symptoms)", 1-"mild", 2-"moderate", 3="severe" and 4= "very severe". Percentage of participants with shift from baseline in PGIS score were reported. A negative shift from baseline in PGIS score indicated Improvement and positive shift from baseline in PGIS score indicated Worsening. The baseline value was defined as the value collected at the time closest to but prior to the randomization.
Time Frame: Baseline, 51.7 months
Population: Analysis population set included in ITT (all randomized) participants with available data for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1: Arm 1A: Erdafitinib 8 mg/9 mg | Cohort 1: Arm 1B: Chemotherapy (Vinflunine 320 mg/m^2 or Docetaxel 75 mg/m^2) | Cohort 2: Arm 2A: Erdafitinib 8 mg/ 9 mg | Cohort 2: Arm 2B: Pembrolizumab 200 mg
Number analyzed (Participants) | 53 | 57 | 104 | 99
Percentage of participants
  -4 Improvement | 0 | 0 | 0 | 0
  -3 | 0 | 0 | 0 | 0
  -2 | 5.7 | 8.8 | 3.8 | 4.0
  -1 | 15.1 | 17.5 | 13.5 | 15.2
  0 No Change | 34.0 | 33.3 | 44.2 | 46.5
  +1 | 30.2 | 26.3 | 20.2 | 17.2
  +2 | 7.5 | 10.5 | 11.5 | 13.1
  +3 | 7.5 | 3.5 | 4.8 | 3.0
  +4 Worsening | 0 | 0 | 1.9 | 1

7. Secondary Outcome: Change From Baseline in Utility Scale of the European Quality of Life-5 Dimensions-5 Levels Questionnaire (EQ-5D-5L)
Description: The EQ-5D-5L was a generic measure of health status. The EQ-5D-5L was a 5-item questionnaire that assessed 5 domains included mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Health utility values generated from the EQ-5D generally range from 0 (a state as bad as being dead) to 1 (full health), with higher scores indicating better QoL. The EQ visual analog scale (VAS) recorded the patient's self-rated health on a VAS, ranged from 0 (worst imaginable health state) to 100 (best imaginable health state), with higher scores indicating better QoL. The baseline value was defined as the value collected at the time closest to but prior to the randomization.
Time Frame: Baseline up to Cycle 11 (each cycle was of 21 days)
Population: Analysis population set included in ITT (all randomized) participants with available data for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Cohort 1: Arm 1A: Erdafitinib 8 mg/9 mg | Cohort 1: Arm 1B: Chemotherapy (Vinflunine 320 mg/m^2 or Docetaxel 75 mg/m^2) | Cohort 2: Arm 2A: Erdafitinib 8 mg/ 9 mg | Cohort 2: Arm 2B: Pembrolizumab 200 mg
Number analyzed (Participants) | 136 | 130 | 175 | 176
Score on a scale | -0.06 (0.023) | -0.06 (0.026) | -0.04 (0.023) | -0.04 (0.024)

8. Secondary Outcome: Change From Baseline in Visual Analog Scale (VAS) of the European Quality of Life-5 Dimensions-5 Levels Questionnaire (EQ-5D-5L)
Description: The EQ-5D-5L was a generic measure of health status. The EQ-5D-5L was a 5-item questionnaire that assessed 5 domains included mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Health utility values generated from the EQ-5D generally range from 0 (a state as bad as being dead) to 1 (full health), with higher scores indicating better QoL. The EQ VAS recorded the patient's self-rated health on a VAS, ranged from 0 (worst imaginable health state) to 100 (best imaginable health state), with higher scores indicating better QoL. The baseline value was defined as the value collected at the time closest to but prior to the randomization.
Time Frame: Baseline up to Cycle 11 (each cycle was of 21 days)
Population: Analysis population set included in ITT (all randomized) participants with available data for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Cohort 1: Arm 1A: Erdafitinib 8 mg/9 mg | Cohort 1: Arm 1B: Chemotherapy (Vinflunine 320 mg/m^2 or Docetaxel 75 mg/m^2) | Cohort 2: Arm 2A: Erdafitinib 8 mg/ 9 mg | Cohort 2: Arm 2B: Pembrolizumab 200 mg
Number analyzed (Participants) | 136 | 130 | 175 | 176
Score on a scale | -0.80 (2.242) | -0.29 (2.626) | -4.16 (2.149) | -2.28 (2.198)

9. Secondary Outcome: Duration of Response (DOR) as Per RECIST Version 1.1
Description: DOR was defined as time from the date of initial documentation of an overall response (CR or PR) to the date of first documented evidence of progressive disease (PD) (or relapse for participants who experience CR) or death. As per RECIST Version 1.1: CR was defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must had reduction in the short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. PD was defined as at least 20% increase in the sum of diameters of measured lesions taking as references the smallest sum of diameters recorded on study (including baseline) and an absolute increase of >=5 mm or appearance of at least 1 new lesion.
Time Frame: From date of first documented response to date of first documented PD or death whichever occurred first (maximum up to 51.7 months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1: Arm 1A: Erdafitinib 8 mg/9 mg | Cohort 1: Arm 1B: Chemotherapy (Vinflunine 320 mg/m^2 or Docetaxel 75 mg/m^2) | Cohort 2: Arm 2A: Erdafitinib 8 mg/ 9 mg | Cohort 2: Arm 2B: Pembrolizumab 200 mg
Number analyzed (Participants) | 67 | 17 | 70 | 38
Months | 4.86 [3.84 to 6.90] | 5.62 [2.79 to 6.01] | 4.67 [3.68 to 6.90] | 15.21 [7.39 to 27.79]

10. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. TEAEs were the events between first dose of study drug and up to 30 days after last dose or before start of new anticancer therapy, whichever occurred first. All TEAEs including serious and non-serious events were reported in this outcome measure.
Time Frame: From start of the treatment (Day 1 Cycle 1) up to 30 days after last dose of study drug or start of subsequent anticancer therapy (maximum up to 51.7 months)
Population: Safety analysis set included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Arm 1A: Erdafitinib 8 mg/9 mg | Cohort 1: Arm 1B: Chemotherapy (Vinflunine 320 mg/m^2 or Docetaxel 75 mg/m^2) | Cohort 2: Arm 2A: Erdafitinib 8 mg/ 9 mg | Cohort 2: Arm 2B: Pembrolizumab 200 mg
Number analyzed (Participants) | 142 | 117 | 173 | 173
Participants | 142 | 114 | 173 | 167

11. Secondary Outcome: Number of Participants With Shift From Baseline Grade Less Than or Equal to (<=) 2 to Grade Greater Than or Equal to (>=) 3 Post-Baseline in Laboratory Parameter: Hematology
Description: Hematology parameters included: hemoglobin, platelet count, white blood cell (WBC) count, and absolute neutrophil count (ANC). According to national cancer institute (NCI)-common terminology criteria for adverse events (CTCAE) version 4.03: Grade 1= mild, Grade 2= moderate, Grade 3= severe, Grade 4= life-threatening, urgent intervention indicated, Grade 5= death related to AE and Grade 0= normal. In this outcome measure number of participants with shifts from baseline (BL) Grade <= 2 to Grade >=3 post-baseline in any of hematology parameters are reported. The baseline value for safety assessment was defined as the value collected at the time closest to, but prior to, the administration of the first dose of study drug. Only those categories in which at least one participant had data were reported in this outcome measure.
Time Frame: From baseline up to 30 days after last dose or start of new anticancer therapy, whichever occurred first (maximum up to 51.7 months)
Population: Safety analysis set included all randomized participants who received at least 1 dose of study drug. Here, 'N' (overall number of participants analyzed) refers to the number of participants evaluable for this outcome measure and 'n' (number analyzed) signifies number of participants evaluable for specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Arm 1A: Erdafitinib 8 mg/9 mg | Cohort 1: Arm 1B: Chemotherapy (Vinflunine 320 mg/m^2 or Docetaxel 75 mg/m^2) | Cohort 2: Arm 2A: Erdafitinib 8 mg/ 9 mg | Cohort 2: Arm 2B: Pembrolizumab 200 mg
Number analyzed (Participants) | 140 | 108 | 171 | 165
Participants
  Anemia: Grade 0 (BL) to Grade 3 (Post BL) | 1 | 2 | 1 | 1
  Anemia: Grade 1 (BL) to Grade 3 (Post BL) | 5 | 6 | 9 | 10
  Anemia: Grade 2 (BL) to Grade 3 (Post BL) | 10 | 4 | 4 | 5
  Hemoglobin Increased: Grade 0 (BL) to Grade 3 (Post BL) | 1 | 0 | 0 | 0
  Neutrophil Count Decreased: Grade 0 (BL) to Grade 3 (Post BL): number analyzed (Participants) | 140 | 108 | 171 | 164
  Neutrophil Count Decreased: Grade 0 (BL) to Grade 3 (Post BL) | 2 | 9 | 0 | 0
  Neutrophil Count Decreased: Grade 0 (BL) to Grade 4 (Post BL): number analyzed (Participants) | 140 | 108 | 171 | 164
  Neutrophil Count Decreased: Grade 0 (BL) to Grade 4 (Post BL) | 0 | 20 | 1 | 1
  Neutrophil Count Decreased: Grade 1 (BL) to Grade 4 (Post BL) | 0 | 1 | 0 | 0
  Platelet Count Decreased: Grade 0 (BL) to Grade 3 (Post BL) | 2 | 1 | 0 | 2
  Platelet Count Decreased: Grade 0 (BL) to Grade 4 (Post BL) | 0 | 1 | 0 | 1
  Platelet Count Decreased: Grade 1 (BL) to Grade 3 (Post BL) | 0 | 0 | 1 | 0
  White Blood Cell Decreased: Grade 0 (BL) to Grade 3 (Post BL) | 0 | 10 | 1 | 2
  White Blood Cell Decreased: Grade 0 (BL) to Grade 4 (Post BL) | 0 | 10 | 1 | 1
  White Blood Cell Decreased: Grade 1 (BL) to Grade 3 (Post BL) | 0 | 2 | 0 | 0

12. Secondary Outcome: Number of Participants With Shift From Baseline Grade <= 2 to Grade >=3 Post-Baseline in Laboratory Parameter: Chemistry
Description: Chemistry parameters included: albumin, alkaline phosphatase (ALP), alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin, chloride, creatinine, bicarbonate, corrected calcium, magnesium, potassium, sodium, serum phosphate, serum parathyroid hormone. According to NCI-CTCAE version 4.03: Grade 1= mild, Grade 2= moderate, Grade 3= severe, Grade 4= life-threatening, urgent intervention indicated, Grade 5= death related to AE and Grade 0= normal. In this outcome measure number of participants with shifts from baseline (BL) Grade <= 2 to Grade >=3 post-baseline in any of chemistry parameters are reported. The baseline value for safety assessment was defined as the value collected at the time closest to, but prior to, the administration of the first dose of study drug. Only those categories in which at least one participant had data were reported in this outcome measure.
Time Frame: as for outcome 11
Population: Safety analysis set included all randomized participants who received at least 1 dose of study drug. Here, 'N' (overall number of participants analyzed) refers to the number of participants evaluable for this outcome measure and 'n' (number analyzed) signifies number of participants evaluable for specified rows. n=0 indicates that no participant was available for the analysis in the respective arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Arm 1A: Erdafitinib 8 mg/9 mg | Cohort 1: Arm 1B: Chemotherapy (Vinflunine 320 mg/m^2 or Docetaxel 75 mg/m^2) | Cohort 2: Arm 2A: Erdafitinib 8 mg/ 9 mg | Cohort 2: Arm 2B: Pembrolizumab 200 mg
Number analyzed (Participants) | 140 | 106 | 173 | 166
Participants
  ALT Increased: Grade 0 (BL) to Grade 3 (Post BL): number analyzed (Participants) | 140 | 105 | 173 | 165
  ALT Increased: Grade 0 (BL) to Grade 3 (Post BL) | 4 | 0 | 4 | 1
  ALT Increased: Grade 0 (BL) to Grade 4 (Post BL): number analyzed (Participants) | 140 | 105 | 173 | 165
  ALT Increased: Grade 0 (BL) to Grade 4 (Post BL) | 0 | 0 | 0 | 2
  ALT Increased: Grade 1 (BL) to Grade 3 (Post BL): number analyzed (Participants) | 140 | 105 | 173 | 165
  ALT Increased: Grade 1 (BL) to Grade 3 (Post BL) | 1 | 1 | 1 | 0
  ALP Increased: Grade 0 (BL) to Grade 3 (Post BL): number analyzed (Participants) | 139 | 104 | 167 | 154
  ALP Increased: Grade 0 (BL) to Grade 3 (Post BL) | 1 | 1 | 1 | 4
  ALP Increased: Grade 1 (BL) to Grade 3 (Post BL): number analyzed (Participants) | 139 | 104 | 167 | 154
  ALP Increased: Grade 1 (BL) to Grade 3 (Post BL) | 5 | 0 | 1 | 2
  ALP Increased: Grade 2 (BL) to Grade 3 (Post BL): number analyzed (Participants) | 139 | 104 | 167 | 154
  ALP Increased: Grade 2 (BL) to Grade 3 (Post BL) | 1 | 1 | 5 | 0
  ALP Increased: Grade 2 (BL) to Grade 4 (Post BL): number analyzed (Participants) | 139 | 104 | 167 | 154
  ALP Increased: Grade 2 (BL) to Grade 4 (Post BL) | 1 | 0 | 0 | 0
  AST Increased: Grade 0 (BL) to Grade 3 (Post BL): number analyzed (Participants) | 139 | 105 | 173 | 164
  AST Increased: Grade 0 (BL) to Grade 3 (Post BL) | 3 | 0 | 1 | 2
  AST Increased: Grade 0 (BL) to Grade 4 (Post BL): number analyzed (Participants) | 139 | 105 | 173 | 164
  AST Increased: Grade 0 (BL) to Grade 4 (Post BL) | 1 | 0 | 0 | 2
  AST Increased: Grade 1 (BL) to Grade 3 (Post BL): number analyzed (Participants) | 139 | 105 | 173 | 164
  AST Increased: Grade 1 (BL) to Grade 3 (Post BL) | 1 | 0 | 2 | 3
  AST Increased: Grade 2 (BL) to Grade 3 (Post BL): number analyzed (Participants) | 0 | 0 | 0 | 164
  AST Increased: Grade 2 (BL) to Grade 3 (Post BL) |  |  |  | 1
  Blood Bilirubin Increased: Grade 0 (BL) to Grade 3 (Post BL): number analyzed (Participants) | 138 | 105 | 173 | 162
  Blood Bilirubin Increased: Grade 0 (BL) to Grade 3 (Post BL) | 1 | 1 | 4 | 1
  Blood Bilirubin Increased: Grade 0 (BL) to Grade 4 (Post BL): number analyzed (Participants) | 138 | 105 | 173 | 162
  Blood Bilirubin Increased: Grade 0 (BL) to Grade 4 (Post BL) | 0 | 0 | 0 | 1
  Blood Bilirubin Increased: Grade 1 (BL) to Grade 3 (Post BL): number analyzed (Participants) | 138 | 0 | 173 | 162
  Blood Bilirubin Increased: Grade 1 (BL) to Grade 3 (Post BL) | 0 |  | 0 | 1
  Blood Bilirubin Increased: Grade 2 (BL) to Grade 3 (Post BL): number analyzed (Participants) | 0 | 105 | 173 | 0
  Blood Bilirubin Increased: Grade 2 (BL) to Grade 3 (Post BL) |  | 0 | 1 |
  Creatinine Increased: Grade 0 (BL) to Grade 3 (Post BL): number analyzed (Participants) | 140 | 105 | 173 | 166
  Creatinine Increased: Grade 0 (BL) to Grade 3 (Post BL) | 0 | 0 | 0 | 3
  Creatinine Increased: Grade 0 (BL) to Grade 4 (Post BL): number analyzed (Participants) | 140 | 105 | 173 | 166
  Creatinine Increased: Grade 0 (BL) to Grade 4 (Post BL) | 0 | 0 | 1 | 0
  Creatinine Increased: Grade 1 (BL) to Grade 3 (Post BL): number analyzed (Participants) | 140 | 105 | 173 | 166
  Creatinine Increased: Grade 1 (BL) to Grade 3 (Post BL) | 1 | 0 | 2 | 1
  Creatinine Increased: Grade 2 (BL) to Grade 3 (Post BL): number analyzed (Participants) | 140 | 105 | 173 | 166
  Creatinine Increased: Grade 2 (BL) to Grade 3 (Post BL) | 2 | 0 | 2 | 3
  Hypercalcemia (Corrected): Grade 0 (BL) to Grade 3 (Post BL): number analyzed (Participants) | 60 | 13 | 34 | 2
  Hypercalcemia (Corrected): Grade 0 (BL) to Grade 3 (Post BL) | 3 | 0 | 0 | 0
  Hypercalcemia (Corrected): Grade 1 (BL) to Grade 3 (Post BL): number analyzed (Participants) | 60 | 13 | 34 | 0
  Hypercalcemia (Corrected): Grade 1 (BL) to Grade 3 (Post BL) | 0 | 0 | 1 |
  Hypercalcemia (Corrected): Grade 1 (BL) to Grade 4 (Post BL): number analyzed (Participants) | 60 | 13 | 34 | 0
  Hypercalcemia (Corrected): Grade 1 (BL) to Grade 4 (Post BL) | 1 | 0 | 1 |
  Hypercalcemia (Corrected): Grade 2 (BL) to Grade 3 (Post BL): number analyzed (Participants) | 60 | 0 | 34 | 2
  Hypercalcemia (Corrected): Grade 2 (BL) to Grade 3 (Post BL) | 0 |  | 0 | 1
  Hyperkalemia: Grade 0 (BL) to Grade 3 (Post BL): number analyzed (Participants) | 140 | 105 | 173 | 166
  Hyperkalemia: Grade 0 (BL) to Grade 3 (Post BL) | 2 | 0 | 5 | 1
  Hyperkalemia: Grade 0 (BL) to Grade 4 (Post BL): number analyzed (Participants) | 140 | 105 | 173 | 166
  Hyperkalemia: Grade 0 (BL) to Grade 4 (Post BL) | 0 | 0 | 0 | 1
  Hyperkalemia: Grade 1 (BL) to Grade 3 (Post BL): number analyzed (Participants) | 140 | 105 | 173 | 166
  Hyperkalemia: Grade 1 (BL) to Grade 3 (Post BL) | 0 | 0 | 1 | 2
  Hyperkalemia: Grade 2 (BL) to Grade 3 (Post BL): number analyzed (Participants) | 140 | 105 | 173 | 166
  Hyperkalemia: Grade 2 (BL) to Grade 3 (Post BL) | 0 | 0 | 1 | 2
  Hypermagnesemia: Grade 0 (BL) to Grade 3 (Post BL): number analyzed (Participants) | 140 | 100 | 164 | 151
  Hypermagnesemia: Grade 0 (BL) to Grade 3 (Post BL) | 3 | 1 | 2 | 1
  Hypermagnesemia: Grade 1 (BL) to Grade 3 (Post BL): number analyzed (Participants) | 0 | 100 | 164 | 151
  Hypermagnesemia: Grade 1 (BL) to Grade 3 (Post BL) |  | 0 | 1 | 1
  Hypernatremia: Grade 0 (BL) to Grade 3 (Post BL): number analyzed (Participants) | 140 | 106 | 165 | 159
  Hypernatremia: Grade 0 (BL) to Grade 3 (Post BL) | 0 | 0 | 0 | 1
  Hyperphosphatemia: Grade 0 (BL) to Grade 3 (Post BL): number analyzed (Participants) | 139 | 30 | 172 | 45
  Hyperphosphatemia: Grade 0 (BL) to Grade 3 (Post BL) | 6 | 0 | 1 | 0
  Hyperphosphatemia: Grade 0 (BL) to Grade 4 (Post BL): number analyzed (Participants) | 139 | 30 | 172 | 45
  Hyperphosphatemia: Grade 0 (BL) to Grade 4 (Post BL) | 1 | 0 | 0 | 0
  Hypoalbuminemia: Grade 0 (BL) to Grade 3 (Post BL): number analyzed (Participants) | 97 | 23 | 62 | 8
  Hypoalbuminemia: Grade 0 (BL) to Grade 3 (Post BL) | 0 | 0 | 0 | 1
  Hypoalbuminemia: Grade 1 (BL) to Grade 3 (Post BL): number analyzed (Participants) | 97 | 23 | 62 | 0
  Hypoalbuminemia: Grade 1 (BL) to Grade 3 (Post BL) | 0 | 1 | 0 |
  Hypocalcemia (Corrected): Grade 0 (BL) to Grade 4 (Post BL): number analyzed (Participants) | 60 | 13 | 34 | 2
  Hypocalcemia (Corrected): Grade 0 (BL) to Grade 4 (Post BL) | 1 | 0 | 0 | 0
  Hypocalcemia (Corrected): Grade 1 (BL) to Grade 3 (Post BL): number analyzed (Participants) | 60 | 13 | 34 | 0
  Hypocalcemia (Corrected): Grade 1 (BL) to Grade 3 (Post BL) | 0 | 0 | 1 |
  Hypokalemia: Grade 0 (BL) to Grade 3 (Post BL): number analyzed (Participants) | 140 | 105 | 173 | 166
  Hypokalemia: Grade 0 (BL) to Grade 3 (Post BL) | 0 | 1 | 4 | 0
  Hypokalemia: Grade 0 (BL) to Grade 4 (Post BL): number analyzed (Participants) | 140 | 105 | 173 | 166
  Hypokalemia: Grade 0 (BL) to Grade 4 (Post BL) | 0 | 0 | 1 | 0
  Hypokalemia: Grade 1 (BL) to Grade 3 (Post BL): number analyzed (Participants) | 0 | 0 | 0 | 166
  Hypokalemia: Grade 1 (BL) to Grade 3 (Post BL) |  |  |  | 1
  Hypokalemia: Grade 2 (BL) to Grade 3 (Post BL): number analyzed (Participants) | 140 | 105 | 173 | 166
  Hypokalemia: Grade 2 (BL) to Grade 3 (Post BL) | 0 | 2 | 0 | 0
  Hypomagnesemia: Grade 1 (BL) to Grade 3 (Post BL): number analyzed (Participants) | 140 | 100 | 164 | 151
  Hypomagnesemia: Grade 1 (BL) to Grade 3 (Post BL) | 0 | 0 | 1 | 1
  Hypomagnesemia: Grade 2 (BL) to Grade 3 (Post BL): number analyzed (Participants) | 0 | 0 | 0 | 151
  Hypomagnesemia: Grade 2 (BL) to Grade 3 (Post BL) |  |  |  | 1
  Hyponatremia: Grade 0 (BL) to Grade 3 (Post BL): number analyzed (Participants) | 140 | 106 | 165 | 159
  Hyponatremia: Grade 0 (BL) to Grade 3 (Post BL) | 14 | 2 | 14 | 4
  Hyponatremia: Grade 0 (BL) to Grade 4 (Post BL): number analyzed (Participants) | 140 | 106 | 165 | 159
  Hyponatremia: Grade 0 (BL) to Grade 4 (Post BL) | 3 | 1 | 1 | 0
  Hyponatremia: Grade 1 (BL) to Grade 3 (Post BL): number analyzed (Participants) | 140 | 106 | 165 | 159
  Hyponatremia: Grade 1 (BL) to Grade 3 (Post BL) | 5 | 4 | 8 | 4
  Hyponatremia: Grade 1 (BL) to Grade 4 (Post BL): number analyzed (Participants) | 140 | 106 | 165 | 159
  Hyponatremia: Grade 1 (BL) to Grade 4 (Post BL) | 0 | 0 | 3 | 1
  Hypophosphatemia: Grade 0 (BL) to Grade 3 (Post BL): number analyzed (Participants) | 139 | 30 | 172 | 45
  Hypophosphatemia: Grade 0 (BL) to Grade 3 (Post BL) | 8 | 1 | 14 | 2
  Hypophosphatemia: Grade 1 (BL) to Grade 3 (Post BL): number analyzed (Participants) | 139 | 0 | 172 | 45
  Hypophosphatemia: Grade 1 (BL) to Grade 3 (Post BL) | 1 |  | 1 | 0
  Hypophosphatemia: Grade 2 (BL) to Grade 3 (Post BL): number analyzed (Participants) | 139 | 30 | 172 | 45
  Hypophosphatemia: Grade 2 (BL) to Grade 3 (Post BL) | 1 | 1 | 1 | 0

13. Secondary Outcome: Number of Participants With Abnormalities in Electrocardiograms (ECG) Parameters
Description: Number of participants with abnormalities in ECG parameters were reported. The ECG variables included heart rate, RR interval, PR interval, QRS interval, QT interval and QT corrected according to Fridericia's formula (QTcF). ECG abnormality criteria include: Heart rate: Low <50 beats per minute (bpm); High > 100 bpm, RR interval: Low < 600 milliseconds (ms); High > 1000 ms, QT interval: High > 500 ms, QTc interval: High > (450 ms for males, 470 ms for females); increase to >500 ms.
Time Frame: Day 1 of Cycle 2 and 4 (Each Cycle 21 days)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Arm 1A: Erdafitinib 8 mg/9 mg | Cohort 1: Arm 1B: Chemotherapy (Vinflunine 320 mg/m^2 or Docetaxel 75 mg/m^2) | Cohort 2: Arm 2A: Erdafitinib 8 mg/ 9 mg | Cohort 2: Arm 2B: Pembrolizumab 200 mg
Number analyzed (Participants) | 130 | 73 | 153 | 150
Participants
  Cycle 2 Day 1 | 31 | 20 | 55 | 47
  Cycle 4 Day 1: number analyzed (Participants) | 104 | 48 | 108 | 109
  Cycle 4 Day 1 | 29 | 13 | 38 | 40

14. Secondary Outcome: Change From Baseline in Vital Signs: Weight
Description: Changes from baseline in vital signs (weight) was reported. The baseline value for safety assessment was defined as the value collected at the time closest to, but prior to, the administration of the first dose of study drug.
Time Frame: Baseline, 51.7 months
Population: Safety analysis set included all randomized participants who received at least 1 dose of study drug. Here, 'N' (overall number of participants analyzed) refers to the number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Cohort 1: Arm 1A: Erdafitinib 8 mg/9 mg | Cohort 1: Arm 1B: Chemotherapy (Vinflunine 320 mg/m^2 or Docetaxel 75 mg/m^2) | Cohort 2: Arm 2A: Erdafitinib 8 mg/ 9 mg | Cohort 2: Arm 2B: Pembrolizumab 200 mg
Number analyzed (Participants) | 76 | 79 | 120 | 115
Kilograms | -5.95 (6.183) | -1.23 (3.580) | -4.13 (5.531) | -1.26 (4.334)

15. Secondary Outcome: Number of Participants With Shift From Baseline to Worst Post-baseline Ophthalmologic Examination: Amsler Grid Test
Description: Number of participants with shift from baseline to worst post-baseline in Amsler grid test was reported. Baseline and post-baseline visit findings included normal, abnormal CS (clinically significant) and abnormal NCS (not clinically significant). Clinical significance was determined by investigator's assessment. The baseline value for safety assessment was defined as the value collected at the time closest to, but prior to, the administration of the first dose of study drug. Only categories in which at least one participant had data for worsening post-baseline measurement was reported.
Time Frame: From baseline up to maximum of 51.7 months
Population: Analysis population set included participants from safety set (SS) with non-missing values for Amsler grid test (AGT) taken at baseline, at least 1 post-baseline visit, and at least 1 visit following the first worst post-baseline value. Due to change in planned analysis, data was collected and analyzed for only Cohort 1 and Cohort 2 Erdafitinib arms.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Arm 1A: Erdafitinib 8 mg/9 mg | Cohort 2: Arm 2A: Erdafitinib 8 mg/ 9 mg
Number analyzed (Participants) | 126 | 165
Participants
  Normal (BL) to Abnormal CS (post-BL) | 20 | 24
  Normal (BL) to Abnormal NCS (post-BL) | 9 | 11
  Abnormal NCS (BL) to Abnormal CS (post-BL) | 5 | 3

16. Secondary Outcome: Number of Participants With Shift From Baseline to Worst Post-baseline Ophthalmologic Examination: Visual Acuity
Description: Number of participants with shift from baseline to worst post-baseline in visual acuity (VA) was reported. Worst post-baseline was defined as the visual acuity value that resulted in the largest change from baseline value for either eye. Baseline value was considered for the eye that reported the worst-post baseline value. Baseline and post-baseline visit visual acuity findings included: <= 20/30, >20/30 to <= 20/40, >20/40 to <= 20/80, >20/80 to <= 20/120, >20/120 to <= 20/160, >20/160 to <= 20/200, >20/200. The baseline value for safety assessment was defined as the value collected at the time closest to, but prior to, the administration of the first dose of study drug. Only categories in which at least one participant had data for worsening in visual acuity from baseline value to worst post-baseline measurement was reported.
Time Frame: From baseline up to maximum of 51.7 months
Population: Analysis set: participants from SS with non-missing values for VA that were convertible to Snellen format taken at BL and at least 1 post BL visit that uses same method. Post BL ophthalmologic examinations were performed only when deemed clinically necessary based on findings of AGT and clinical assessment, or at regular intervals as deemed necessary by screening ophthalmologist. Due to change in planned analysis, data was collected and analyzed for only Cohort 1 and Cohort 2 Erdafitinib arms.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Arm 1A: Erdafitinib 8 mg/9 mg | Cohort 2: Arm 2A: Erdafitinib 8 mg/ 9 mg
Number analyzed (Participants) | 41 | 46
Participants
  <= 20/30 (BL) To >20/30 to <= 20/40 (Post BL) | 10 | 11
  <= 20/30 (BL) To >20/40 to <= 20/80 (Post BL) | 2 | 5
  <= 20/30 (BL) To >20/80 to <= 20/120 (Post BL) | 2 | 1
  <= 20/30 (BL) To >20/120 to <= 20/160 (Post BL) | 1 | 1
  <= 20/30 (BL) To >20/160 to <= 20/200 (Post BL) | 5 | 1
  <= 20/30 (BL) To >20/200 (post BL) | 0 | 1
  >20/30 to <= 20/40 (BL) To >20/40 to <= 20/80 (Post BL) | 0 | 4
  >20/30 to <= 20/40 (BL) To >20/160 to <= 20/200 (Post BL) | 0 | 1

17. Secondary Outcome: Number of Participants With Shift From Baseline to Worst Post-baseline Ophthalmologic Examination: Optical Coherence Tomography: Subretinal Fluid
Description: Number of participants with shift from baseline to worst post-baseline in optical coherence tomography for subretinal fluid was reported. At the baseline visit, findings may have been absent or present/visible. At all post-baseline visits, findings were compared to baseline and results may have been increased, decreased, stable or resolved. The baseline value for safety assessment was defined as the value collected at the time closest to, but prior to, the administration of the first dose of study drug. Only category (shift from absent at baseline to increased at post-baseline) in which at least one participant had data for worsening post-baseline measurement was reported.
Time Frame: From baseline up to maximum of 51.7 months
Population: Analysis population set: participants from safety set with non-missing values for the subretinal fluid at baseline and at least 1 post-baseline visit. Post-baseline ophthalmologic examinations were performed only when deemed clinically necessary based on the findings of the Amsler grid tests and clinical assessment, or at regular intervals as deemed necessary by the screening ophthalmologist. Due to change in planned analysis, data was collected and analyzed for Cohort 1 Erdafitinib arm only.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Arm 1A: Erdafitinib 8 mg/9 mg
Number analyzed (Participants) | 39
Participants | 26

18. Secondary Outcome: Number of Participants With Shift From Baseline to Worst Post-baseline Ophthalmologic Examination: Optical Coherence Tomography: Retinal Pigment Epithelium (RPE) Elevation
Description: Number of participants with shift from baseline to worst post-baseline in optical coherence tomography for RPE elevation was reported. At the baseline visit, findings may have been absent or present/visible. At all post-baseline visits, findings were compared to baseline and results may have been increased, decreased, stable or resolved. The baseline value for safety assessment was defined as the value collected at the time closest to, but prior to, the administration of the first dose of study drug. Only categories in which at least one participant had data for worsening post-baseline measurement was reported.
Time Frame: From baseline up to maximum of 51.7 months
Population: Analysis population set: participants from safety set with non-missing values for the RPE elevation at baseline and at least 1 post-baseline visit. Post-baseline ophthalmologic examinations were performed only when deemed clinically necessary based on the findings of the Amsler grid tests and clinical assessment, or at regular intervals as deemed necessary by the screening ophthalmologist. Due to change in planned analysis, data was collected and analyzed for Cohort 1 Erdafitinib arm only.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Arm 1A: Erdafitinib 8 mg/9 mg
Number analyzed (Participants) | 38
Participants
  Absent (BL) to Increased (Post BL) | 4
  Present/visible (BL) to Increased (Post BL) | 2

19. Secondary Outcome: Number of Participants With Shift From Baseline to Worst Post-baseline Ophthalmologic Examination: Slit Lamp Biomicroscopy: Retinal Assessment
Description: Number of participants with shift from baseline to worst post-baseline in slit lamp biomicroscopy examination for retinal assessment was reported. Baseline and post-baseline visit findings included normal, abnormal CS and abnormal NCS. Clinical significance was determined by investigator's assessment. The baseline value for safety assessment was defined as the value collected at the time closest to, but prior to, the administration of the first dose of study drug. Only categories in which at least one participant had data for worsening post-baseline measurement was reported.
Time Frame: From baseline up to maximum of 51.7 months
Population: Analysis population set: participants from SS with non-missing values for retinal assessments at baseline and at least 1 post-baseline visit. Post-baseline ophthalmologic examinations were performed only when deemed clinically necessary based on the findings of the Amsler grid tests and clinical assessment, or at regular intervals as deemed necessary by screening ophthalmologist. Due to change in planned analysis, data was collected and analyzed for only Cohort 1 and Cohort 2 Erdafitinib arms.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Arm 1A: Erdafitinib 8 mg/9 mg | Cohort 2: Arm 2A: Erdafitinib 8 mg/ 9 mg
Number analyzed (Participants) | 39 | 47
Participants
  Normal (BL) to Abnormal CS (post-BL) | 3 | 4
  Normal (BL) to Abnormal NCS (post-BL) | 5 | 6
  Abnormal NCS (BL) to Abnormal CS (post-BL) | 1 | 0

20. Secondary Outcome: Oral Clearance (CL/F) of Erdafitinib
Description: Clearance was a measure of the rate at which a drug was metabolized or eliminated by normal biological processes.
Time Frame: Day 14 of Cycle 1, Day 1 of Cycle 2: pre-dose and 2-4 hours post-dose (each cycle was of 21 days)
Population: Pharmacokinetic-evaluable analysis set included all randomized participants who received at least 1 dose of erdafitinib and had at least 1 evaluable pharmacokinetic sample obtained posttreatment. Here 'N' (overall number of participants analyzed) refers to the number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Liter per hour
Arm/Group | Cohort 1: Arm 1A: Erdafitinib 8 mg/9 mg | Cohort 2: Arm 2A: Erdafitinib 8 mg/ 9 mg
Number analyzed (Participants) | 126 | 149
Liter per hour | NA (NA) — Here, NA signifies that data could not be analyzed as due to sparse PK sampling, the data were insufficient to derive CL/F using non-compartmental analysis (NCA) method. | NA (NA) — Here, NA signifies that data could not be analyzed as due to sparse PK sampling, the data were insufficient to derive CL/F using NCA method.

21. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Time 't' (AUC[0-t]) of Erdafitinib
Description: Area under the plasma concentration time-curve from time zero to the time t (AUC[0-t]) was reported.
Time Frame: Day 14 of Cycle 1, Day 1 of Cycle 2: pre-dose and 2-4 hours post-dose (each cycle is of 21 days)
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Nanogram hour per milliliter
Arm/Group | Cohort 1: Arm 1A: Erdafitinib 8 mg/9 mg | Cohort 2: Arm 2A: Erdafitinib 8 mg/ 9 mg
Number analyzed (Participants) | 126 | 149
Nanogram hour per milliliter | NA (NA) — Here, NA signifies that data could not be analyzed as due to sparse PK sampling, the data were insufficient to derive AUC using NCA method. | NA (NA) — Here, NA signifies that data could not be analyzed as due to sparse PK sampling, the data were insufficient to derive AUC using NCA method.

ADVERSE EVENTS:
Time Frame: All-cause mortality: From randomization (3 days prior to Cycle 1 Day 1) up to maximum of 51.7 months; serious AEs and other AEs: From Day 1 Cycle 1 up to maximum of 51.7 months
Description: Serious/other AEs: Safety analysis set. All-cause mortality: ITT population (all randomized). The study was to evaluate efficacy of erdafitinib versus standard chemotherapy chosen at site level by investigators. Regardless of which chemotherapy was chosen by investigator (docetaxel/vinflunine), AEs were collected and analyzed collectively for chemotherapy arm (Vinflunine 320 mg/m^2 or Docetaxel 75 mg/m^2; Arm 1B). Per plan safety was analyzed per intervention.
Arm/Group | Cohort 1: Arm 1A: Erdafitinib 8 mg/9 mg | Cohort 1: Arm 1B: Chemotherapy (Vinflunine 320 mg/m^2 or Docetaxel 75 mg/m^2) | Cohort 2: Arm 2A: Erdafitinib 8 mg/ 9 mg | Cohort 2: Arm 2B: Pembrolizumab 200 mg
All-Cause Mortality (participants affected / at risk) | 91/143 | 90/135 | 141/175 | 131/176
Serious Adverse Events (participants affected / at risk) | 63/142 | 50/117 | 69/173 | 81/173
Other Adverse Events (participants affected / at risk) | 141/142 | 104/117 | 173/173 | 157/173
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Arm 1A: Erdafitinib 8 mg/9 mg (N=142) | Cohort 1: Arm 1B: Chemotherapy (Vinflunine 320 mg/m^2 or Docetaxel 75 mg/m^2) (N=117) | Cohort 2: Arm 2A: Erdafitinib 8 mg/ 9 mg (N=173) | Cohort 2: Arm 2B: Pembrolizumab 200 mg (N=173)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 1 | 3
Bone Marrow Failure (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Febrile Bone Marrow Aplasia (Blood and lymphatic system disorders) | 0 | 4 | 0 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 8 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0
Myelosuppression (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 3 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0
Acute Coronary Syndrome (Cardiac disorders) | 1 | 0 | 0 | 0
Acute Myocardial Infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Angina Pectoris (Cardiac disorders) | 0 | 1 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac Arrest (Cardiac disorders) | 1 | 0 | 0 | 1
Cardiac Tamponade (Cardiac disorders) | 1 | 0 | 0 | 0
Cardio-Respiratory Arrest (Cardiac disorders) | 1 | 0 | 1 | 0
Sinus Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Stress Cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 | 0
Supraventricular Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Vestibular Disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Adrenal Insufficiency (Endocrine disorders) | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 1 | 0 | 0 | 0
Detachment of Retinal Pigment Epithelium (Eye disorders) | 2 | 0 | 2 | 0
Keratitis (Eye disorders) | 0 | 0 | 2 | 0
Serous Retinal Detachment (Eye disorders) | 0 | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 2 | 3 | 0
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Colo-Urethral Fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Duodenal Ulcer Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Enterovesical Fistula (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastric Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Gastrointestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal Perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 1 | 1 | 1
Inguinal Hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Intestinal Ischaemia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0 | 6 | 2
Intestinal Perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Large Intestine Perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Mechanical Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 2 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 1 | 2 | 0
Subileus (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Asthenia (General disorders) | 2 | 0 | 0 | 3
Condition Aggravated (General disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 1
General Physical Health Deterioration (General disorders) | 1 | 3 | 2 | 4
Malaise (General disorders) | 0 | 0 | 1 | 0
Multiple Organ Dysfunction Syndrome (General disorders) | 0 | 0 | 1 | 1
Non-Cardiac Chest Pain (General disorders) | 0 | 1 | 0 | 1
Pain (General disorders) | 0 | 1 | 0 | 0
Performance Status Decreased (General disorders) | 0 | 0 | 0 | 1
Precancerous Condition (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 2 | 3 | 1 | 2
Sudden Death (General disorders) | 2 | 0 | 0 | 0
Biliary Obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 1 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Hepatic Function Abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hepatobiliary Disease (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Abdominal Infection (Infections and infestations) | 1 | 1 | 0 | 0
Abdominal Sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Anal Abscess (Infections and infestations) | 1 | 0 | 0 | 0
Appendicitis Perforated (Infections and infestations) | 0 | 0 | 1 | 0
Atypical Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 2 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Clostridium Difficile Infection (Infections and infestations) | 0 | 1 | 0 | 0
Covid-19 (Infections and infestations) | 1 | 0 | 0 | 1
Covid-19 Pneumonia (Infections and infestations) | 0 | 0 | 2 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1
Device Related Infection (Infections and infestations) | 0 | 1 | 0 | 0
Endocarditis (Infections and infestations) | 0 | 0 | 1 | 0
Kidney Infection (Infections and infestations) | 1 | 0 | 0 | 0
Large Intestine Infection (Infections and infestations) | 0 | 1 | 0 | 0
Localised Infection (Infections and infestations) | 0 | 0 | 1 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0 | 0
Perinephric Abscess (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 2 | 1 | 5
Pneumonia Aspiration (Infections and infestations) | 2 | 0 | 0 | 0
Pneumonia Necrotising (Infections and infestations) | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 2 | 3 | 3
Pyelonephritis Acute (Infections and infestations) | 1 | 0 | 1 | 0
Pyelonephritis Chronic (Infections and infestations) | 0 | 0 | 0 | 1
Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 2 | 0 | 1 | 2
Septic Shock (Infections and infestations) | 0 | 2 | 3 | 1
Soft Tissue Infection (Infections and infestations) | 0 | 0 | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0 | 0
Urinary Tract Candidiasis (Infections and infestations) | 0 | 1 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 7 | 3 | 6 | 9
Urinary Tract Infection Enterococcal (Infections and infestations) | 0 | 1 | 0 | 0
Urinary Tract Infection Pseudomonal (Infections and infestations) | 1 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 1 | 2 | 1
Viral Infection (Infections and infestations) | 0 | 0 | 1 | 0
Compression Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Toxicity to Various Agents (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Urinary Tract Stoma Complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Urostomy Complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Blood Creatinine Increased (Investigations) | 1 | 0 | 0 | 1
Urine Output Decreased (Investigations) | 0 | 0 | 1 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 0 | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 1 | 0 | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 1 | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Bladder Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 2 | 1
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Hepatic Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Metastases to Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Cerebral Ischaemia (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 0 | 0 | 1
Cognitive Disorder (Nervous system disorders) | 0 | 0 | 1 | 0
Dysarthria (Nervous system disorders) | 1 | 0 | 0 | 0
Generalised Tonic-Clonic Seizure (Nervous system disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Paralysis (Nervous system disorders) | 1 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0 | 0
Spinal Cord Compression (Nervous system disorders) | 0 | 0 | 0 | 1
Device Occlusion (Product Issues) | 0 | 0 | 0 | 1
Confusional State (Psychiatric disorders) | 1 | 0 | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 3 | 0 | 6 | 6
Bladder Dysfunction (Renal and urinary disorders) | 0 | 0 | 0 | 1
Bladder Obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 1
Bladder Perforation (Renal and urinary disorders) | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 5 | 1 | 3 | 5
Hydronephrosis (Renal and urinary disorders) | 2 | 0 | 0 | 2
Micturition Urgency (Renal and urinary disorders) | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal Colic (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal Failure (Renal and urinary disorders) | 2 | 0 | 2 | 2
Renal Impairment (Renal and urinary disorders) | 0 | 0 | 0 | 1
Ureteric Obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 3
Ureteric Stenosis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urethral Haemorrhage (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary Incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary Retention (Renal and urinary disorders) | 1 | 1 | 2 | 2
Urinary Tract Obstruction (Renal and urinary disorders) | 2 | 1 | 2 | 0
Pelvic Pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
Prostatitis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 2 | 4
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 4
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 2
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Haemorrhage Subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Nail Dystrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Onycholysis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Toxic Skin Eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Catheter Placement (Surgical and medical procedures) | 0 | 1 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 1 | 1
Dry Gangrene (Vascular disorders) | 1 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 1
Embolism Venous (Vascular disorders) | 0 | 0 | 0 | 1
Extremity Necrosis (Vascular disorders) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 2 | 1 | 0 | 0
Peripheral Artery Aneurysm (Vascular disorders) | 0 | 0 | 0 | 1
Peripheral Ischaemia (Vascular disorders) | 1 | 0 | 1 | 0
Vascular Calcification (Vascular disorders) | 1 | 0 | 0 | 0
Venous Thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Arm 1A: Erdafitinib 8 mg/9 mg (N=142) | Cohort 1: Arm 1B: Chemotherapy (Vinflunine 320 mg/m^2 or Docetaxel 75 mg/m^2) (N=117) | Cohort 2: Arm 2A: Erdafitinib 8 mg/ 9 mg (N=173) | Cohort 2: Arm 2B: Pembrolizumab 200 mg (N=173)
Anaemia (Blood and lymphatic system disorders) | 40 | 39 | 51 | 44
Leukopenia (Blood and lymphatic system disorders) | 1 | 15 | 5 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 24 | 3 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 9 | 13 | 12
Hyperparathyroidism (Endocrine disorders) | 8 | 0 | 4 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 1 | 0 | 9
Hypothyroidism (Endocrine disorders) | 2 | 1 | 0 | 19
Chorioretinopathy (Eye disorders) | 10 | 0 | 12 | 0
Detachment of Retinal Pigment Epithelium (Eye disorders) | 8 | 0 | 8 | 0
Dry Eye (Eye disorders) | 28 | 2 | 22 | 2
Keratitis (Eye disorders) | 9 | 1 | 8 | 0
Lacrimation Increased (Eye disorders) | 12 | 1 | 17 | 0
Vision Blurred (Eye disorders) | 14 | 0 | 10 | 1
Visual Impairment (Eye disorders) | 4 | 1 | 9 | 1
Xerophthalmia (Eye disorders) | 8 | 1 | 9 | 1
Abdominal Pain (Gastrointestinal disorders) | 11 | 8 | 20 | 10
Abdominal Pain Upper (Gastrointestinal disorders) | 4 | 1 | 11 | 5
Constipation (Gastrointestinal disorders) | 44 | 32 | 40 | 38
Diarrhoea (Gastrointestinal disorders) | 90 | 22 | 92 | 23
Dry Mouth (Gastrointestinal disorders) | 61 | 4 | 63 | 8
Dyspepsia (Gastrointestinal disorders) | 6 | 2 | 12 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 8 | 4 | 2 | 1
Mouth Ulceration (Gastrointestinal disorders) | 9 | 2 | 4 | 0
Nausea (Gastrointestinal disorders) | 20 | 27 | 28 | 19
Stomatitis (Gastrointestinal disorders) | 74 | 17 | 83 | 6
Vomiting (Gastrointestinal disorders) | 14 | 15 | 24 | 9
Asthenia (General disorders) | 22 | 29 | 48 | 37
Fatigue (General disorders) | 22 | 23 | 29 | 24
Oedema Peripheral (General disorders) | 9 | 17 | 15 | 19
Pyrexia (General disorders) | 21 | 15 | 12 | 20
Conjunctivitis (Infections and infestations) | 14 | 0 | 17 | 3
Covid-19 (Infections and infestations) | 12 | 6 | 3 | 5
Nail Infection (Infections and infestations) | 8 | 0 | 2 | 0
Paronychia (Infections and infestations) | 20 | 0 | 12 | 3
Urinary Tract Infection (Infections and infestations) | 13 | 7 | 19 | 31
Alanine Aminotransferase Increased (Investigations) | 39 | 5 | 28 | 13
Aspartate Aminotransferase Increased (Investigations) | 31 | 3 | 29 | 14
Blood Alkaline Phosphatase Increased (Investigations) | 18 | 3 | 17 | 8
Blood Creatinine Increased (Investigations) | 20 | 9 | 27 | 12
Weight Decreased (Investigations) | 33 | 3 | 28 | 7
Decreased Appetite (Metabolism and nutrition disorders) | 40 | 25 | 57 | 21
Hypercalcaemia (Metabolism and nutrition disorders) | 11 | 1 | 7 | 8
Hyperkalaemia (Metabolism and nutrition disorders) | 9 | 3 | 13 | 7
Hyperphosphataemia (Metabolism and nutrition disorders) | 117 | 0 | 134 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 | 5 | 9 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 8 | 3 | 2 | 5
Hyponatraemia (Metabolism and nutrition disorders) | 17 | 3 | 24 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 | 9 | 21 | 14
Back Pain (Musculoskeletal and connective tissue disorders) | 11 | 11 | 19 | 22
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 11 | 3 | 4
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 14 | 6 | 19 | 8
Dizziness (Nervous system disorders) | 4 | 6 | 3 | 5
Dysgeusia (Nervous system disorders) | 43 | 8 | 42 | 1
Headache (Nervous system disorders) | 4 | 7 | 4 | 6
Peripheral Sensory Neuropathy (Nervous system disorders) | 5 | 9 | 6 | 2
Insomnia (Psychiatric disorders) | 6 | 8 | 2 | 6
Haematuria (Renal and urinary disorders) | 15 | 11 | 22 | 20
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 10 | 5 | 17
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 7 | 8 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 18 | 4 | 19 | 1
Nasal Dryness (Respiratory, thoracic and mediastinal disorders) | 6 | 0 | 9 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 37 | 28 | 31 | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 34 | 5 | 43 | 9
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 9 | 0
Nail Discolouration (Skin and subcutaneous tissue disorders) | 25 | 2 | 29 | 0
Nail Disorder (Skin and subcutaneous tissue disorders) | 20 | 2 | 11 | 2
Nail Dystrophy (Skin and subcutaneous tissue disorders) | 15 | 0 | 20 | 0
Nail Ridging (Skin and subcutaneous tissue disorders) | 8 | 1 | 1 | 0
Onycholysis (Skin and subcutaneous tissue disorders) | 36 | 1 | 42 | 0
Onychomadesis (Skin and subcutaneous tissue disorders) | 29 | 3 | 15 | 0
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 44 | 2 | 38 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 2 | 7 | 24
Rash (Skin and subcutaneous tissue disorders) | 7 | 5 | 6 | 15
Xeroderma (Skin and subcutaneous tissue disorders) | 4 | 1 | 9 | 0
Hypertension (Vascular disorders) | 1 | 3 | 4 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2023-01-20): https://cdn.clinicaltrials.gov/large-docs/04/NCT03390504/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-24): https://cdn.clinicaltrials.gov/large-docs/04/NCT03390504/SAP_001.pdf